CLINICAL TRIAL: NCT01516307
Title: A Double-blind, Randomized Trial of Active Immunotherapy With Globo H-KLH (OPT-822) in Subjects With Metastatic Breast Cancer
Brief Title: Trial of Active Immunotherapy With Globo H-KLH (OPT-822) in Metastatic Breast Cancer Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPT-822-001
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OPT-822/OPT-821 (30 μg/100 μg) and Cyclophosphamide (Experimental): Patients will be randomized 2:1 to receive OPT-822/OPT-821(30 μg/100 μg) plus Cyclophosphamide IV (300mg/m2).
  Interventions: Biological: OPT-822/OPT-821(30 μg/100 μg); Drug: Cyclophosphamide
- Phosphate Buffer Saline (PBS) and Cyclophosphamide (Placebo Comparator): Patients will receive Phosphate Buffer Saline (PBS) plus Cyclophosphamide IV (300mg/m2).
  Interventions: Biological: Phosphate Buffer Saline (PBS); Drug: Cyclophosphamide

INTERVENTIONS:
Biological: OPT-822/OPT-821(30 μg/100 μg) — Subcutaneously on week 1, 2, 3, 5, 9, 13, 17, 25, and 37. OPT-822 and OPT-821 are combined at time of injection.
  Arms: OPT-822/OPT-821 (30 μg/100 μg) and Cyclophosphamide
Biological: Phosphate Buffer Saline (PBS) — Subcutaneously on week 1, 2, 3, 5, 9, 13, 17, 25, and 37.
  Arms: Phosphate Buffer Saline (PBS) and Cyclophosphamide
Drug: Cyclophosphamide — Subcutaneously on week 1, 2, 3, 5, 9, 13, 17, 25, and 37.

SUMMARY:
The purpose of this study is to compare active immunotherapy (OPT-822/OPT-821) with PBS in combination with low dose cyclophosphamide, in post-treated metastatic breast cancer subjects with stable disease or response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects ≥ 21 years of age with histological or cytological diagnosis of breast carcinoma.
* Subjects with metastatic breast cancer who have achieved stable disease (SD), partial response (PR), or complete response (CR) after at least 1 regimen of anticancer therapy (i.e. chemotherapy or target therapy, either alone or in any combination). Involvement of supraclavicular lymph node is considered metastasis.
* Subjects must have recovered from toxicities of prior therapies. (i.e. CTCAE ≤ grade 2).
* Performance status: ECOG ≤ 1 and life expectancy ≥ 3 months.
* Organ Function Requirements - Subjects must have adequate organ functions as defined below:

  * AST/ALT ≤ 3X ULN (upper limit of normal)
  * AST/ALT ≤ 5X ULN [with underlying Liver Metastasis]
  * Total Bilirubin ≤ 2.0 X ULN
  * Serum Creatinine ≤ 1.5X ULN
  * ANC ≥ 1500 /μL
  * Platelets > 100,000/μL
  * No Symptomatic Congestive Heart Failure (Ejection Fraction EF ≥ 50%)
* Ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.
* All positive or negative ER (estrogen receptor), PR (progesterone receptor), and HER-2 subjects are eligible for this study.
* However, subjects who are HER-2 positive and responsive to anti-HER-2 therapy (e.g. Herceptin), are encouraged to remain on anti-HER-2 therapy and not enroll in this trial.
* Subjects who desire to enroll in this study and for whom anti-HER-2 therapy is not available or contraindicated, may be eligible to enroll in this trial.
* In countries where continuous anti-HER2 therapy is considered standard of care for HER-2 positive metastatic disease, HER-2 positive subjects are not eligible.
* Women of childbearing potential must be willing to implement adequate contraception during the study. An adequate method of contraception will be at the investigator's discretion.

Exclusion Criteria:

* Subjects are pregnant or breast-feeding at entry.
* Subjects with more than 2 events of disease progression after the development of metastatic breast cancer.
* Subjects who are currently receiving any other concomitant anticancer therapy with the EXCEPTION of bisphosphonates and hormone therapy.

  * During the study period, subjects using hormonal therapy and bisphosphonates should maintain a constant dose and should not change existing regimen.
  * However, if a change in hormonal therapy is indicated, e.g. due to intolerable adverse effects, the regimen may be modified but change should be minimized thereafter.
* Subjects with metastasis limited to the bone only are excluded. However, subjects with current metastasis limited to the bone only and with a history of distant metastasis are eligible. Subjects with current metastasis limited to the bone only and with current breast tissue lesion are eligible.
* Subjects who have any history of other malignancy (except non-melanoma skin carcinoma and carcinoma-in-situ of the uterine cervix) within 5 years of study entry.
* Subjects with splenectomy.
* Subjects with HIV infection.
* Subjects with any major autoimmune diseases or autoimmune disorders requiring systemic iv/oral steroids or immunosuppressive or immunomodulatory therapies.

  * e.g. Type 1 juvenile onset diabetes mellitus, antibody positive for rheumatoid arthritis, Grave's disease, Hashimoto's thyroiditis, lupus, scleroderma, systemic vasculitis, hemolytic anemia, immune mediated thrombocytopenia, etc
  * Autoimmune disorders confined to the skin (e.g. psoriasis) are eligible, and topical steroids are allowed for the treatment of such skin disorders.
* Subjects with any known uncontrolled inter-current illness including ongoing or active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with any of the following MEDICATIONS within 4 weeks prior to randomization:

  * Anti-neoplastic agents
  * Immunotherapy [mAbs, Interferons, Cytokines (except GCSF)]
  * Immunosuppressants (e.g. Cyclosporin, Rapamycin, Tacrolimus, Rituximab, Alemtuzumab, Natalizumab, etc.).
  * Another investigational drug
* Subjects with pleural effusions and/or ascites, due to malignancy, requiring paracentesis every 2 weeks or more frequently.
* Subjects with any known severe allergies (e.g. anaphylaxis) to any active or inactive ingredients in the study drugs.
* Subjects with bladder inflammation and urinary outflow obstruction.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2011-12; Primary Completion 2016-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Progression or up to 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Locations (43):
- United States (13):
  - The University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - St. Jude Heritage Healthcare, Virginia K. Crosson Cancer Center, Fullerton, California
  - University of California, San Diego (UCSD), La Jolla, California
  - University of California, Irvine (UCI), Orange, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - University of California, Los Angeles (UCLA), Santa Monica, California
  - Memorial Regional Hospital, Hollywood, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Weill Cornell Medical College, New York, New York
  - Hope Women's Cancer Center, Asheville, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- UNIMED Medical Institute, Hong Kong, China
- India (2):
  - HCG, Bangalore Institute of Oncology, Bengaluru
  - Curie Manavata Cancer Centre, Mumbai
- South Korea (11):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Inha University Hospital, Chungcheongbuk-Do
  - National Cancer Center, Chungcheongbuk-Do
  - Kyungpook National University Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital ,, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Seoul
- Taiwan (16):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital-KS, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital -Linkou, Linkou District
  - Mackay Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital-Taipei, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Shuang-Ho Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CS, Yu AL, Tseng LM, Chow LWC, Hou MF, Hurvitz SA, Schwab RB, L Murray J, Chang HK, Chang HT, Chen SC, Kim SB, Hung JT, Ueng SH, Lee SH, Chen CC, Rugo HS. Globo H-KLH vaccine adagloxad simolenin (OBI-822)/OBI-821 in patients with metastatic breast cancer: phase II randomized, placebo-controlled study. J Immunother Cancer. 2020 Jul;8(2):e000342. doi: 10.1136/jitc-2019-000342. PMID 32718986